CLINICAL TRIAL: NCT02333110
Title: Spatially Fractionated Radiation (SFR) Therapy as Palliative Radiation for Patients With Advanced and Symptomatic Tumors
Brief Title: GRID Therapy as Palliative Radiation for Patients With Advanced and Symptomatic Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Te Vuong, Director, Radiation-oncology department, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-161
Record Dates: First submitted 2014-12-22; First posted 2015-01-07 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Patients With Symptomatic or Bulky Tumors (More Than 8 cm) or With Tumors Resistant to Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GRID radiation therapy (Experimental): A single dose of 15-20Gys of spatially fractionated radiation therapy
  Interventions: Radiation: spatially fractionated radiation therapy

INTERVENTIONS:
Radiation: spatially fractionated radiation therapy — A single dose of 15-20Gys of spatially fractionated radiation therapy
  Other Names: GRID radiation therapy

SUMMARY:
Palliative radiation therapy represents 40% of the on-going radiation at the Jewish General Hospital. In a traditional palliative radiation treatment to bulky or radioresistant tumors, radiotherapy schema varies from 24 to 30 Gys given in 3 to 10 fractions, depending on the tumor size, tumor location and tumor pathology. However, for many patients this treatment involves considerable toxicity, travel and time spent at the hospital. Spatially fractionated radiation (SFR) is an alternative technique that consists in delivering one single treatment, given through a grid containing holes. The present study is proposing to validate SFR as a safe and effective mean to palliate patients with symptomatic bulky tumors (more than 8 cm) or with tumors known to be resistant to radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically or cytologically confirmed malignancy. All malignant histologies/cytologies are eligible.
* Patient with bulky tumor (larger than 8cm), or with a tumor known to be resistant to radiation (eg. Melanoma, hypernephroma, sarcoma), or with a tumor previously irradiated with a palliative intent requiring more than 1 fraction of radiation
* Patient planned to undergo palliative radiation therapy treatments to one of the following 5 sites: extremities, neck, chest, abdomen and pelvis
* WHO performance status of 0-2
* Aged 18 years or older
* Ability to sign and understand an informed consent form

Exclusion Criteria:

* Potentially curable patient
* Previous palliative radiation with hypofractionation
* Tumor located near the spinal cord or in the brain
* Pregnant or nursing woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Symptom relief, as measured using the CTCAE grading system (v4.0) and pain questionnaire | 3 months post treatment

SECONDARY OUTCOMES:
Acute toxicity of treatment, as measured using the CTCAE grading system (v4.0) | 1 week
Long-term toxicity of treatment, as measured using the CTCAE grading system (v4.0) | 3, 6, 9, 12 months
Cost-effectiveness, as measured by evaluating the cost of the procedure per patient and the efficacy of treatment with regards to symptom relief and tumor response | 3 months
Tumor response, measured on CT-scan | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Te Vuong, MD, Principal Investigator — Sir Mortimer Jewish General Hospital
Locations (1):
- Sir Mortimer Jewish General Hospital, Montreal, Quebec, Canada